CLINICAL TRIAL: NCT04016181
Title: The Edinburgh Lung Fibrosis Molecular Endotyping (ELFMEN) Study
Acronym: ELFMEN
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 07/S1102/20; 2007/R/RES/02 (Other: University of Edinburgh and NHS Lothian)
Record Dates: First submitted 2019-03-29; First posted 2019-07-11 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease; Asbestosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial; Asbestosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Serum EDTA blood Bronchoalveolar lavage (fluid and cells) Lung biopsy (fresh and formalin fixed)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To prospectively study novel blood and lung biomarkers of disease activity in patients with IPF and other interstitial lung disease with the aims of prognostic modelling and disease clustering

DETAILED DESCRIPTION:
BACKGROUND

Idiopathic pulmonary fibrosis (IPF) is a progressive form of lung scarring for which there is no proven treatment. Steroids and other potentially toxic drugs are often used but their efficacy is uncertain. The management of patients with IPF is particularly complex because firstly there are a number of closely related fibrosing lung conditions that 'look' like IPF but in which the prognosis is generally better and which more often respond to steroids and secondly even within the group of patients with IPF, there is a variability in the rate of progression so that it is hard to provide individual patients with a reasonable estimate of prognosis.

Currently the best the investigators can offer patients with IPF or other fibrotic interstitial lung disease is serial measurement of lung function over time and observation of decline. The uncertainty regarding disease prognosis and progression in a given patient is hugely unsettling for both the individual and the clinician. A far more powerful tool would be a measurement or 'biomarker' of disease activity that one could monitor from the time of diagnosis and throughout the illness and which predicted for decline in lung function or poor prognosis. This biomarker (or biomarkers) might include molecules associated with inflammation and scarring in blood or in lung fluid, new more sensitive measures of lung function (e.g. the six-minute walking test) or novel non-invasive imaging methods. Once established, a robust biomarker would serve several important functions including:

1. Prognostication of individuals with IPF and other fibrotic ILDs
2. Identifying targets for potential new therapies in IPF and other fibtroic ILDs
3. A marker of disease response to drugs used in therapeutic trials in IPF and other fibrotic ILDs.
4. A means of distinguishing definite IPF from other closely related conditions;

   AIMS To prospectively study novel blood and lung biomarkers of disease activity in patients with IPF and other interstitial lung disease

   STUDY DESIGN Inclusion criteria Patients attending or referred to the Edinburgh Royal Infirmary and the Western General Hospital lung fibrosis clinics with a diagnosis of definite or probable idiopathic pulmonary fibrosis. For comparison patients with other idiopathic interstitial pneumonias, hypersensitivity pneumonitis, asbestosis or interstitial lung disease associated with connective tissue diseases will also be recruited since these conditions often have a similar clinical presentation to IPF but a more variable prognosis. All clinical details for these patients are already being collated in a REC-approved clinical database (REC 06/S0703/53). Patients aged 18 through 99 years, inclusive.

   Exclusion criteria and restrictions Candidates not a suitable for enrolment or unlikely to comply with the requirements of this study, in the opinion of the investigator, will be excluded.

   The biomarkers will include assays that test the activity of circulating blood inflammatory cells in laboratory conditions. A relatively large volume of blood (up to 80ml a time) is required to purify sufficient numbers of these inflammatory cells for use in laboratory studies. It is anticipated however that as data is gathered, subsequent experiments can be refined such that less blood is required.

   No more than 320ml of blood over a 12 month period will be taken from any study participant for research purposes. No more than 100ml of blood over a twelve month period will be taken from any study participant with a moderate or severe anaemia, defined as a haemoglobin >10% below lower limit of normal. Anaemia is not a recognised complication of idiopathic pulmonary fibrosis.

   Participants that are deemed unsuitable for bronchoscopy, based on established national and local guidelines, will be excluded from this aspect of the study.

   WHAT WILL HAPPEN TO THE RESEARCH PARTICIPANTS
   * indicates routine clinical investigations performed on all patients with IPF or other interstitial lung disease • indicates study investigations, some of which are may performed as part of routine clinical care

   Within 1 month of presentation or recruitment to the study participants will undergo:
   * Blood samples for routine biochemistry, haematology, auto-immune screen and other clinically relevant tests
   * Full lung function tests and incremental walking test
   * HRCT scan •Bronchoalveolar lavage (BAL) - note that this may be performed for clinical diagnostic indications in many patients with suspected IPF.

     * Blood sample for biomarkers (average 40ml, not >80ml)

   At 3 months following recruitment participants will undergo:

   *Blood sample for biomarkers (average 40ml, not >80ml)

   At 6 months following recruitment participants will undergo:

   •Blood sample for biomarkers (average 40ml, not >80ml)

   At 9 months following recruitment participants will undergo:

   •Blood sample for biomarkers (average 40ml, not >80ml)

   At 12 months following recruitment participants will undergo:

   •Bronchoalveolar lavage

   •Blood sample for biomarkers (average 40ml, not >80ml)

   Thereafter repeated every 6 months for up to 3 years, participants will undergo:

   •Blood sample for biomarkers (average 40ml, not >80ml)

   In patients that have a lung biopsy for clinical indications, resected lung tissue that is deemed not critical to the diagnostic process by pathologist i.e. excess fresh tissue, will be used for research purposes. To ensure this is safely achieved, excess lung tissue will stored and not used for research until the pathologist has confirmed that available material is sufficient for clinical purposes. In practice, this means a sample of fresh tissue form the 'staple' margins of the resected specimen. Formalin fixed archived tissue from subjects will be included for use in this study. This protocol was used in a previous ethically approved study (09/S1101/52, Molecular markers of hypoxia, cell injury and fibrosis in lung tissue. This study ended 31/3/15 having collected 40 consecutive fresh lung fibrosis specimens without incident.

   STUDY OUTCOMES (see endpoints) Identification of prognostics biomarkers in all entities of ILD including IPF that define disease progression and death Identification of novel disease entity clusters define by clinical, imaging and molecular features

ELIGIBILITY:
Inclusion Criteria:

* patients with interstitial lung disease attending the Edinburgh Lung Fibrosis service

Exclusion Criteria:

* candidates not a suitable for enrolment or unlikely to comply with the requirements of this study, in the opinion of the investigator, will be excluded.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with all entities of interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2007-06-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to death (all cause) | 15 years
  Biomarkers that are associated with increased all-cause mortality

SECONDARY OUTCOMES:
Rate of decline in vital capacity | 15 years
  Biomarkers that are associated with increased rate of decline in vital capacity (VC)
Time to death (lung-related) | 15 years
  Biomarkers that are associated with increased lung-related mortality
Rate of decline in TLCO | 15 years
  Biomarkers that predict rate of change in gas transfer (TLCO)

OTHER OUTCOMES:
Identification of novel disease clusters | 15 years
  Identification of discrete disease entities based on clinical, imaging and molecular data
Time to oxygen prescription | 15 years
  Biomarkers that are associated with reduced time to prescription of long term oxygen

IPD SHARING:
Plan to Share IPD: Undecided
sharing of individual participant data will be determined on a case-by-case basis contingent of data security governance

REFERENCES:
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625